CLINICAL TRIAL: NCT06411834
Title: Mapping Patient Decision-making in Thyroid Cancer: Improving Decision Outcomes Through Ethnographic Decision Modeling
Brief Title: Mapping Patient Decision-making in Thyroid Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, James Wu, MD, Assistant Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-001913
Record Dates: First submitted 2023-06-09; First posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Thyroid Cancer
Keywords: decision-making
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decision Navigation Tool (Experimental): Patients will be asked to complete a decision navigation tool that helps them identify and rank key decision criteria. Then we will use a predictive model to inform patients which initial treatment options similar patients have made, and which choices lead to high satisfaction and low regret.
  Interventions: Behavioral: Decision navigation tool
- Usual care (No Intervention): Patients will undergo usual care

INTERVENTIONS:
Behavioral: Decision navigation tool — An electronic, interactive form that guides patients through the major factors that influence their decision-making in thyroid cancer
  Arms: Decision Navigation Tool

SUMMARY:
The incidence of thyroid cancer has exploded in the past 5 decades, with a roughly three-fold increase since 1995. Fortunately, many new cases are small, early-stage thyroid cancers. The American Thyroid Association guidelines state that patients with papillary thyroid cancers less than 4 cm can choose either thyroid lobectomy or total thyroidectomy. However, it is unclear why patients will sometimes choose more aggressive treatments that carry additional operative risk when a less aggressive option is available. When investigators examined thyroid specialists' recommendations for thyroid cancer treatment, investigators found significant variation between physicians' risk estimates and their treatment recommendations. This illustrated that patients may receive inconsistent counseling regarding their diagnosis and treatment options from different providers. Worse yet, other studies have shown that patients often do not perceive a choice in their treatment. When patients undergo treatments that do not align with their own priorities and values, they may experience regret and low satisfaction. Decision aids have been shown to help patients feel more educated about their options but have not had an effect on their treatment choice, decision regret, or satisfaction.

The aim of this study is to use an ethnographic approach to map the patient decision-making process and develop a Decision Navigation Tool to improve decision outcomes for thyroid cancer patients. An ethnographic approach seeks to understand the social norms, culture, and context that influence these decisions. Investigators will do so in 3 phases: 1) elicit patient decision criteria in selecting initial treatment for thyroid cancer, 2) construction and validation of decision-tree model for initial treatment of thyroid cancer, and 3) pilot randomized controlled trial of a Decision Navigation Tool. To construct the decision model, investigators will recruit a diverse sample of patients with varying age, gender, race/ethnicity, and operative and cancer outcomes. The Decision Navigation Tool will highlight patients' values and priorities and empower them to select a treatment aligned with their preferences. This study will provide important insights into the patient experience of decision-making in thyroid cancer and test the feasibility of a future multi-center large-scale clinical trial of a Decision Navigation Tool to improve decision outcomes.

DETAILED DESCRIPTION:
The incidence of thyroid cancer has exploded in the past 5 decades, with a roughly three-fold increase since 1995. Fortunately, many new cases are small, early-stage thyroid cancers. The American Thyroid Association guidelines state that patients with papillary thyroid cancers less than 4 cm can choose either thyroid lobectomy or total thyroidectomy. However, it is unclear why patients will sometimes choose more aggressive treatments that carry additional operative risk when a less aggressive option is available. When investigators examined thyroid specialists' recommendations for thyroid cancer treatment, investigators found significant variation between physicians' risk estimates and their treatment recommendations. This illustrated that patients may receive inconsistent counseling regarding their diagnosis and treatment options from different providers. Worse yet, other studies have shown that patients often do not perceive a choice in their treatment. When patients undergo treatments that do not align with their own priorities and values, they may experience regret and low satisfaction. Decision aids have been shown to help patients feel more educated about their options but have not had an effect on their treatment choice, decision regret, or satisfaction.

The aim of this study is to use an ethnographic approach to map the patient decision-making process and develop a Decision Navigation Tool to improve decision outcomes for thyroid cancer patients. An ethnographic approach seeks to understand the social norms, culture, and context that influence these decisions. Investigators will do so in 3 phases: 1) elicit patient decision criteria in selecting initial treatment for thyroid cancer, 2) construction and validation of decision-tree model for initial treatment of thyroid cancer, and 3) pilot randomized controlled trial of a Decision Navigation Tool. To construct the decision model, investigators will recruit a diverse sample of patients with varying age, gender, race/ethnicity, and operative and cancer outcomes. The Decision Navigation Tool will highlight patients' values and priorities and empower them to select a treatment aligned with their preferences. This study will provide important insights into the patient experience of decision-making in thyroid cancer and test the feasibility of a future multi-center large-scale clinical trial of a Decision Navigation Tool to improve decision outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Newly diagnosed or suspected thyroid cancer

Exclusion Criteria:

* Strong indication for total thyroidectomy
* tumor size >4 cm
* nodal or distant metastases
* evidence of extrathyroidal extension
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Decision satisfaction | 1 year postoperative
  University of Ottawa Decisional Conflict Scale
Decision satisfaction | Immediately postoperative
  University of Ottawa Decisional Conflict Scale
Decision satisfaction | Two weeks postoperative
  University of Ottawa Decisional Conflict Scale
Decision regret | 1 year postoperative
  University of Ottawa Decisional Conflict Scale
Decision regret | immediately postoperative
  University of Ottawa Decisional Conflict Scale
Decision regret | two weeks postoperative postoperative
  University of Ottawa Decisional Conflict Scale
Rate of guideline concordant care vs guideline discordant care | During study period of 12 months

IPD SHARING:
Plan to Share IPD: No